CLINICAL TRIAL: NCT03306797
Title: Hand Rehabilitation With Music Therapy Technique (Sonification) and Leap Motion Controller in Stroke Patients
Brief Title: Music Therapy for Rehabilitation in Stroke Patients
Acronym: SONICHAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituti Clinici Scientifici Maugeri SpA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2088 CE
Record Dates: First submitted 2017-08-04; First posted 2017-10-11 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Stroke; Hand Injuries
Keywords: Music therapy; Sonification technique; Rehabilitation
MeSH Terms: conditions — Stroke; Hand Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SONICHAND (Experimental): The intervention is similar to the standard protocol (15 minutes of warm-up plus 20 minute of training) but involves the sonification of the exercises (4 weeks, daily)
  Interventions: Device: SONICHAND
- STANDARD REHAB (Other): The rehabilitative standard intervention (Occupational Therapy) consists of 15 minutes of warm-up exercises plus a 20 minutes training for 4 weeks (daily)
  Interventions: Other: STANDARD REHAB

INTERVENTIONS:
Other: STANDARD REHAB — The rehabilitative standard intervention (Occupational Therapy) consists of 15 minutes of warm-up exercises plus a 20 minutes training with at least 6 exercises selected from:
  wrist
  * ulnarization radialization
  * prono-supination
  * horizontal flexion-extension
  * vertical flexion-extension hand
  * grasping
  * pinching
  * extensors
  * interosseous shoulder-elbow
  * vertical flexion-extension
  * push forward
  Arms: STANDARD REHAB
Device: SONICHAND — The intervention is similar to the standard protocol (15 minutes of warm-up plus 20 minute of training) but involves the sonification of the exercises selected from the list. The Leap Motion Controller is managed with an ad-hoc developed application that is able to associate the movements with a 4 notes arpeggio or with a modulated texture.
  With the first mode the movement produces and modulates an harmonic progression built on the consecutive grades of the major scale played as ascending and descending arpeggio with also a volume crescendo and decrescendo.
  With the second mode, the movement modulates the volume and the low-pass cutoff frequency of a synthetic texture.
  Arms: SONICHAND

SUMMARY:
The study uses a specific hand tracking sensor (Leap Motion Controller) to catch the movements of the arm combined with proper pre-defined musical patterns (sonification) in a neurologic music therapy perspective. The aim of the experiment is to verify the efficacy of sonification technique (compared to usual care) in the hand rehabilitation of patients with stroke.

DETAILED DESCRIPTION:
Introduction:

Every year in Italy occur over than 200.000 new stroke cases. The virtual and augmented reality offers a valid support to the rehabilitation program by providing objectives parameters for the patient evaluation, accelerating the motor recovery process and enhancing the motor performance after the discharge. This study uses a specific hand tracking sensor (Leap Motion Controller) to catch the movements of the arm combined with proper pre-defined musical patterns (sonification) in a neurologic music therapy perspective.

In addition to its use in relational contexts, in fact, music therapy is widely used in the field of rehabilitation, and in particular in the neuromotor rehabilitation, due to the impact of the sound, as well as on paralimbic and limbic areas, the areas of the brain involved in the movements (motor cortex, supplementary motor area, cerebellum, basal ganglia, etc.).

Recent studies uses sonification for the rehabilitation of the upper limbs assuming a replacement of the proprioceptive aspects damaged by the disease thanks to the audio-motor feedback. This study, furthermore, exploits the specificities of the Leap Motion Controller and the peculiarities of the sound stimuli that accompany the arm movement without requiring cognitive tasks.

Objectives:

* To verify through a randomized controlled trial and a suitable motor assessment the efficacy of the rehabilitation of the hand in patients with stroke using the "sonification" technique
* To verify whether the "sonification" technique reduces the fatigue and the pain perceived during rehabilitation
* Assess the impact of "sonification" technique on patients quality of life

Materials and Methods:

In this randomized controlled trial 66 patients with stroke will be recruited and allocated in 2 groups. The control group will be undergone to a 35 minutes standard daily rehabilitation treatment lasting 4 weeks. The experimental group will be undergone to an analogue treatment based on 15 minutes of standard rehabilitation and 20 minutes of exercises with sonification. Randomisation will be centralized for the four Units involved in the study.

The intervention will be assessed in blind at the baseline (T0), at the mid-treatment period (T1 = 2 weeks), at the end of the treatment (T2 = 4 weeks), and at a follow-up point (T3 = 8 weeks).

The following assessment tools will be used:

* Fugl-Meyer Motor Assessment Scale
* Box and Block Test
* Modified Ashworth Scale
* Visual Analogue Scale (VAS)
* Numerical Pain Rating Scale
* McGill Quality of Life

At T0, T1, T2 and T3 some motion parameters will be recorded and monitored by the Leap Motion Controller to evaluate possible changes in the movements execution.

Statistics:

The Intention-To-Treat (ITT) population will be considered for the analysis. An unpaired Student's t test on the pre (T0)-post treatment (T2) differences will be used to assess the primary endpoint. Longitudinal trends over time will be assessed through repeated measures analysis of variance. Other analyses will be available in the statistical analysis plan.

ELIGIBILITY:
Inclusion Criteria:

* 40-85 years old
* ischemic lesion in one hemisphere (hemiplegia / hemiparesis right or left)
* Mini Mental State Examination > 24 onset acute event not later than 180 days prior to study entry

Exclusion Criteria:

* Dated lesions beyond 6 months from onset
* Multiple or bilateral lesions
* Mini Mental State Examination <24
* Presence of neglect
* Previous or concomitant disabling diseases for upper limb function (Eg: Parkinson's disease, multiple sclerosis, shoulder's periarthritis, Dupuytren's disease, etc.)
* Previous rehabilitative treatments with music

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2017-03-28 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Motor Assessment Scale | 4 weeks
  Primary endpoint of the study is given by the measurement of proximal and distal upper limb motor skills assessed by the Fugl-Meyer Motor Assessment Scale. The primary endpoint will be assessed by comparing the variation between T0 and T2 of the scale scores above mentioned in the experimental and control groups.

SECONDARY OUTCOMES:
Box and Block Test (BBT) | up to 8 weeks
  Assessment of unilateral gross manual dexterity
Modified Ashworth Scale | up to 8 weeks
  Measurement of spasticity
Visual Analogue Scale (VAS) | up to 8 weeks
  Evaluation of perceived fatigue
Numerical Pain Rating Scale (NPRS) | up to 8 weeks
  Assessment of pain intensity
McGill Quality of Life | up to 8 weeks
  Assessment of Quality of Life

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (4):
  - ICS Maugeri, Nervi Institute, Genoa, Genova
  - ICS Maugeri, Montescano Institute, Montescano, Pavia
  - ICS Maugeri, Pavia Institute, Pavia
  - Fondazione Santa Lucia IRCCS, Rome

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Altenmuller E, Marco-Pallares J, Munte TF, Schneider S. Neural reorganization underlies improvement in stroke-induced motor dysfunction by music-supported therapy. Ann N Y Acad Sci. 2009 Jul;1169:395-405. doi: 10.1111/j.1749-6632.2009.04580.x. PMID 19673814
- [Background] Bangert M, Altenmuller EO. Mapping perception to action in piano practice: a longitudinal DC-EEG study. BMC Neurosci. 2003 Oct 15;4:26. doi: 10.1186/1471-2202-4-26. PMID 14575529
- [Background] Bangert M, Peschel T, Schlaug G, Rotte M, Drescher D, Hinrichs H, Heinze HJ, Altenmuller E. Shared networks for auditory and motor processing in professional pianists: evidence from fMRI conjunction. Neuroimage. 2006 Apr 15;30(3):917-26. doi: 10.1016/j.neuroimage.2005.10.044. Epub 2005 Dec 27. PMID 16380270
- [Background] Baumann S, Koeneke S, Schmidt CF, Meyer M, Lutz K, Jancke L. A network for audio-motor coordination in skilled pianists and non-musicians. Brain Res. 2007 Aug 3;1161:65-78. doi: 10.1016/j.brainres.2007.05.045. Epub 2007 Jun 4. PMID 17603027
- [Background] Cha Y, Kim Y, Hwang S, Chung Y. Intensive gait training with rhythmic auditory stimulation in individuals with chronic hemiparetic stroke: a pilot randomized controlled study. NeuroRehabilitation. 2014;35(4):681-8. doi: 10.3233/NRE-141182. PMID 25318784
- [Background] Chen P, Lai CKY, Chung RCK, Ng SSM. The Jacket Test for assessing people with chronic stroke. Disabil Rehabil. 2017 Dec;39(25):2577-2583. doi: 10.1080/09638288.2016.1236413. Epub 2016 Oct 28. PMID 27793076
- [Background] Chong HJ, Han SJ, Kim YJ, Park HY, Kim SJ. Relationship between output from MIDI-keyboard playing and hand function assessments on affected hand after stroke. NeuroRehabilitation. 2014;35(4):673-80. doi: 10.3233/NRE-141166. PMID 25318775
- [Background] Conklyn D, Novak E, Boissy A, Bethoux F, Chemali K. The effects of modified melodic intonation therapy on nonfluent aphasia: a pilot study. J Speech Lang Hear Res. 2012 Oct;55(5):1463-71. doi: 10.1044/1092-4388(2012/11-0105). Epub 2012 Mar 12. PMID 22411278
- [Background] Desrosiers J, Bravo G, Hebert R, Dutil E, Mercier L. Validation of the Box and Block Test as a measure of dexterity of elderly people: reliability, validity, and norms studies. Arch Phys Med Rehabil. 1994 Jul;75(7):751-5. PMID 8024419
- [Background] Hayden R, Clair AA, Johnson G, Otto D. The effect of rhythmic auditory stimulation (RAS) on physical therapy outcomes for patients in gait training following stroke: a feasibility study. Int J Neurosci. 2009;119(12):2183-95. doi: 10.3109/00207450903152609. PMID 19916847
- [Background] Huskisson EC. Measurement of pain. Lancet. 1974 Nov 9;2(7889):1127-31. doi: 10.1016/s0140-6736(74)90884-8. No abstract available. PMID 4139420
- [Background] Kim SJ, Koh I. The effects of music on pain perception of stroke patients during upper extremity joint exercises. J Music Ther. 2005 Spring;42(1):81-92. doi: 10.1093/jmt/42.1.81. PMID 15839735
- [Background] Kim DS, Park YG, Choi JH, Im SH, Jung KJ, Cha YA, Jung CO, Yoon YH. Effects of music therapy on mood in stroke patients. Yonsei Med J. 2011 Nov;52(6):977-81. doi: 10.3349/ymj.2011.52.6.977. PMID 22028163
- [Background] Kim SJ, Jo U. Study of accent-based music speech protocol development for improving voice problems in stroke patients with mixed dysarthria. NeuroRehabilitation. 2013;32(1):185-90. doi: 10.3233/NRE-130835. PMID 23422471
- [Background] Iosa M, Morone G, Fusco A, Castagnoli M, Fusco FR, Pratesi L, Paolucci S. Leap motion controlled videogame-based therapy for rehabilitation of elderly patients with subacute stroke: a feasibility pilot study. Top Stroke Rehabil. 2015 Aug;22(4):306-16. doi: 10.1179/1074935714Z.0000000036. Epub 2015 Feb 25. PMID 26258456
- [Background] Jun EM, Roh YH, Kim MJ. The effect of music-movement therapy on physical and psychological states of stroke patients. J Clin Nurs. 2013 Jan;22(1-2):22-31. doi: 10.1111/j.1365-2702.2012.04243.x. Epub 2012 Sep 17. PMID 22978325
- [Background] Gregson JM, Leathley MJ, Moore AP, Smith TL, Sharma AK, Watkins CL. Reliability of measurements of muscle tone and muscle power in stroke patients. Age Ageing. 2000 May;29(3):223-8. doi: 10.1093/ageing/29.3.223. PMID 10855904
- [Background] Lim KB, Kim YK, Lee HJ, Yoo J, Hwang JY, Kim JA, Kim SK. The therapeutic effect of neurologic music therapy and speech language therapy in post-stroke aphasic patients. Ann Rehabil Med. 2013 Aug;37(4):556-62. doi: 10.5535/arm.2013.37.4.556. Epub 2013 Aug 26. PMID 24020037
- [Background] Magee WL, Davidson JW. The effect of music therapy on mood states in neurological patients: a pilot study. J Music Ther. 2002 Spring;39(1):20-9. doi: 10.1093/jmt/39.1.20. PMID 12015809
- [Background] Meyer M, Elmer S, Baumann S, Jancke L. Short-term plasticity in the auditory system: differential neural responses to perception and imagery of speech and music. Restor Neurol Neurosci. 2007;25(3-4):411-31. PMID 17943016
- [Background] Purdie H, Hamilton S, Baldwin S. Music therapy: facilitating behavioural and psychological change in people with stroke--a pilot study. Int J Rehabil Res. 1997 Sep;20(3):325-7. No abstract available. PMID 9331582
- [Background] Sarkamo T, Tervaniemi M, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M. Music listening enhances cognitive recovery and mood after middle cerebral artery stroke. Brain. 2008 Mar;131(Pt 3):866-76. doi: 10.1093/brain/awn013. PMID 18287122
- [Background] Sarkamo T, Pihko E, Laitinen S, Forsblom A, Soinila S, Mikkonen M, Autti T, Silvennoinen HM, Erkkila J, Laine M, Peretz I, Hietanen M, Tervaniemi M. Music and speech listening enhance the recovery of early sensory processing after stroke. J Cogn Neurosci. 2010 Dec;22(12):2716-27. doi: 10.1162/jocn.2009.21376. PMID 19925203
- [Background] Schlaug G. Part VI introduction: listening to and making music facilitates brain recovery processes. Ann N Y Acad Sci. 2009 Jul;1169:372-3. doi: 10.1111/j.1749-6632.2009.04869.x. No abstract available. PMID 19673811
- [Background] Schneider S, Schonle PW, Altenmuller E, Munte TF. Using musical instruments to improve motor skill recovery following a stroke. J Neurol. 2007 Oct;254(10):1339-46. doi: 10.1007/s00415-006-0523-2. Epub 2007 Jan 27. PMID 17260171
- [Background] Scholz DS, Rohde S, Nikmaram N, Bruckner HP, Grossbach M, Rollnik JD, Altenmuller EO. Sonification of Arm Movements in Stroke Rehabilitation - A Novel Approach in Neurologic Music Therapy. Front Neurol. 2016 Jun 30;7:106. doi: 10.3389/fneur.2016.00106. eCollection 2016. PMID 27445970
- [Background] Scholz DS, Rhode S, Grossbach M, Rollnik J, Altenmuller E. Moving with music for stroke rehabilitation: a sonification feasibility study. Ann N Y Acad Sci. 2015 Mar;1337:69-76. doi: 10.1111/nyas.12691. PMID 25773619
- [Background] Scholz DS, Wu L, Pirzer J, Schneider J, Rollnik JD, Grossbach M, Altenmuller EO. Sonification as a possible stroke rehabilitation strategy. Front Neurosci. 2014 Oct 20;8:332. doi: 10.3389/fnins.2014.00332. eCollection 2014. PMID 25368548
- [Background] Sguazzin C, Giorgi I, Alesii A, Fini M. Italian validation of the McGill Quality of Life Questionnaire (MQOL-It). G Ital Med Lav Ergon. 2010 Jul-Sep;32(3 Suppl B):B58-62. PMID 21299077
- [Background] Smeragliuolo AH, Hill NJ, Disla L, Putrino D. Validation of the Leap Motion Controller using markered motion capture technology. J Biomech. 2016 Jun 14;49(9):1742-1750. doi: 10.1016/j.jbiomech.2016.04.006. Epub 2016 Apr 8. PMID 27102160
- [Background] Suh JH, Han SJ, Jeon SY, Kim HJ, Lee JE, Yoon TS, Chong HJ. Effect of rhythmic auditory stimulation on gait and balance in hemiplegic stroke patients. NeuroRehabilitation. 2014;34(1):193-9. doi: 10.3233/NRE-131008. PMID 24284453
- [Background] Tamplin J, Baker FA, Jones B, Way A, Lee S. 'Stroke a Chord': the effect of singing in a community choir on mood and social engagement for people living with aphasia following a stroke. NeuroRehabilitation. 2013;32(4):929-41. doi: 10.3233/NRE-130916. PMID 23867418
- [Background] Thaut MH, McIntosh GC, Rice RR. Rhythmic facilitation of gait training in hemiparetic stroke rehabilitation. J Neurol Sci. 1997 Oct 22;151(2):207-12. doi: 10.1016/s0022-510x(97)00146-9. PMID 9349677
- [Background] Thaut MH, Leins AK, Rice RR, Argstatter H, Kenyon GP, McIntosh GC, Bolay HV, Fetter M. Rhythmic auditory stimulation improves gait more than NDT/Bobath training in near-ambulatory patients early poststroke: a single-blind, randomized trial. Neurorehabil Neural Repair. 2007 Sep-Oct;21(5):455-9. doi: 10.1177/1545968307300523. Epub 2007 Apr 10. PMID 17426347
- [Background] Tung JY, Lulic T, Gonzalez DA, Tran J, Dickerson CR, Roy EA. Evaluation of a portable markerless finger position capture device: accuracy of the Leap Motion controller in healthy adults. Physiol Meas. 2015 May;36(5):1025-35. doi: 10.1088/0967-3334/36/5/1025. Epub 2015 Apr 22. PMID 25902961
- [Background] van Delden AL, Peper CL, Nienhuys KN, Zijp NI, Beek PJ, Kwakkel G. Unilateral versus bilateral upper limb training after stroke: the Upper Limb Training After Stroke clinical trial. Stroke. 2013 Sep;44(9):2613-6. doi: 10.1161/STROKEAHA.113.001969. Epub 2013 Jul 18. PMID 23868279
- [Background] van Wijck F, Knox D, Dodds C, Cassidy G, Alexander G, MacDonald R. Making music after stroke: using musical activities to enhance arm function. Ann N Y Acad Sci. 2012 Apr;1252:305-11. doi: 10.1111/j.1749-6632.2011.06403.x. PMID 22524372
- [Background] Villeneuve M, Penhune V, Lamontagne A. A piano training program to improve manual dexterity and upper extremity function in chronic stroke survivors. Front Hum Neurosci. 2014 Aug 22;8:662. doi: 10.3389/fnhum.2014.00662. eCollection 2014. PMID 25202258
- [Background] Weichert F, Bachmann D, Rudak B, Fisseler D. Analysis of the accuracy and robustness of the leap motion controller. Sensors (Basel). 2013 May 14;13(5):6380-93. doi: 10.3390/s130506380. PMID 23673678
- [Background] Wittwer JE, Webster KE, Hill K. Rhythmic auditory cueing to improve walking in patients with neurological conditions other than Parkinson's disease--what is the evidence? Disabil Rehabil. 2013 Jan;35(2):164-76. doi: 10.3109/09638288.2012.690495. Epub 2012 Jun 8. PMID 22681598